CLINICAL TRIAL: NCT00003771
Title: Protocol for Randomized Clinical Study Concerning Hormonal Replacement Therapy (HRT) After Previous Radical Breast Cancer Treatment
Brief Title: Hormone Replacement Therapy and the Risk of Breast Cancer Recurrence in Women With Previous Early Stage Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regional Oncologic Center (Other)
Collaborators: Scandinavian Breast Group (Other); ETOP IBCSG Partners Foundation (Network); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000066897; ROC-HABITS; EORTC-10992; IBCSG-17-98; SBG-HABITS; EU-98077
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-07

CONDITIONS: Breast Cancer; Menopausal Symptoms
Keywords: menopausal symptoms; stage I breast cancer; stage II breast cancer; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ | interventions — Estradiol; Norethindrone Acetate

INTERVENTIONS:
Biological: therapeutic estradiol
Drug: norethindrone acetate

SUMMARY:
RATIONALE: Hormone replacement therapy is effective for relieving symptoms of menopause. It is not yet known if hormone replacement therapy increases the risk of breast cancer recurrence in women previously treated for early stage breast cancer.

PURPOSE: Randomized phase III trial to determine the risk of breast cancer recurrence in women with previous early stage breast cancer who are receiving hormone replacement therapy for menopause symptoms.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the safety of hormone replacement therapy, in terms of risk of recurrence, in women with previously treated, nonrecurrent stage 0-II breast cancer.
* Compare this regimen vs non-hormonal symptomatic treatment, in terms of quality of life and risk of death, in this patient population.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified by center, prior hormone replacement therapy before diagnosis, and concurrent tamoxifen therapy. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive one of the following: Women with an intact uterus whose last menstrual bleeding has occurred within 2 years receive continuous oral cyclic estradiol-norethindrone combination comprising estradiol only on days 1-12, estradiol plus norethindrone on days 13-22, and then estradiol only on days 22-28. Women with an intact uterus whose last menstrual bleeding occurred more than 2 years prior to study receive continuous daily oral estradiol-norethindrone combination. Women who have had a hysterectomy receive continuous daily oral estradiol only.
* Arm II: Patients receive one or more non-hormonal therapies (e.g., clonidine, beta blockers, psychological support, physical exercise, acupuncture).

Treatment in both arms continues for 2 years in the absence of disease progression. Patients may continue their randomized treatment regimen at the discretion of the treating physician.

Quality of life is assessed 3 times during the study and then every two years thereafter. Gynecological health is assessed at 3 months, 6 months, and one year during the study and then annually for at least 5 years. Breast cancer is assessed every 6 months for 3 years and then annually thereafter or at the discretion of the treating physician.

PROJECTED ACCRUAL: A total of 1,300 patients will be accrued for this study within 5-6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of stage 0-II breast cancer with no more than 4 involved axillary nodes if nodal status and number of nodes investigated is known
* No current evidence of disease
* Hormone receptor status:

  * Positive, negative, or unknown

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Menopausal or perimenopausal

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No active liver disease

Renal:

* Not specified

Cardiovascular:

* No prior or concurrent deep vein thrombosis
* No hereditary traits for deep vein thrombosis
* No prior or concurrent cerebral stroke
* No prior or concurrent coronary disease

Other:

* No prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No porphyria
* No other serious disease that would prevent compliance or greatly limit life expectancy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* Prior hormone replacement therapy (HRT) allowed if stopped no more than 4 weeks after breast cancer diagnosis and at least 3 months prior to study
* No prior HRT initiated after breast cancer diagnosis
* No concurrent hormonal therapy for breast cancer except tamoxifen or toremifene

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No prior randomization into trials comparing effects of chemotherapy and bilateral oophorectomy in premenopausal women

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 1997-09; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Holmberg, MD, PhD, Study Chair — Uppsala University Hospital; Jonas Bergh, MD, PhD, Study Chair — Karolinska Institutet; C. Rageth, MD, PD, Study Chair — Breast Center; Janusz Jaskiewicz, MD, Study Chair — Maria Sklodowska-Curie National Research Institute of Oncology
Locations (6):
- Helsinki University Central Hospital, Helsinki, Finland
- Norwegian Radium Hospital, Oslo, Norway
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Sweden (2):
  - Karolinska Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- Breast Center, Zurich, Switzerland

REFERENCES:
- [Background] Brincat M, Muscat Baron Y, Ciantar E. Hormone replacement in women with breast cancer: the HABITS study. Endocrine. 2004 Aug;24(3):255-7. doi: 10.1385/endo:24:3:255. PMID 15542894
- [Result] Holmberg L, Iversen OE, Rudenstam CM, Hammar M, Kumpulainen E, Jaskiewicz J, Jassem J, Dobaczewska D, Fjosne HE, Peralta O, Arriagada R, Holmqvist M, Maenpaa J; HABITS Study Group. Increased risk of recurrence after hormone replacement therapy in breast cancer survivors. J Natl Cancer Inst. 2008 Apr 2;100(7):475-82. doi: 10.1093/jnci/djn058. Epub 2008 Mar 25. PMID 18364505
- [Result] Holmberg L, Anderson H; HABITS steering and data monitoring committees. HABITS (hormonal replacement therapy after breast cancer--is it safe?), a randomised comparison: trial stopped. Lancet. 2004 Feb 7;363(9407):453-5. doi: 10.1016/S0140-6736(04)15493-7. PMID 14962527